CLINICAL TRIAL: NCT05983822
Title: Robotic Hand Rehabilitation in Stroke Patients
Brief Title: Robotic Hand Rehabilitation
Acronym: RoHa-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, GIOVANNINI SILVIA, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0000052/23
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Spasticity as Sequela of Stroke; Upper Limb
Keywords: Stroke; Robotic rehabilitation; Upper limb
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (GA) (Experimental): The experimental group (GA) will perform specific rehabilitation for the recovery of hand function using the end-effector robot Amadeo® (Tyromotion, Austria) 3 times a week, for 4 weeks (12 total sessions), for 45 minutes of treatment in addition to conventional treatment. In particular, the technological rehabilitation performed using the robot will mostly aim at improving finger mobility and strength, and flexion-extension exercises will be proposed in passive, active assisted and active mode, exercises for improving strength and muscle tone.
  Interventions: Device: Technological Group
- Conventional Group (GC) (Active Comparator): GC patients will undergo conventional rehabilitation treatment only, using the main rehabilitation methods (e.g. neurocognitive theory, progressive neuromuscular facilitation, etc.).
  Interventions: Device: Technological Group; Other: Conventional Treatment

INTERVENTIONS:
Device: Technological Group — Specific rehabilitation for the recovery of hand function using the end-effector robot
  Other Names: Amadeo® (Tyromotion, Austria)
Other: Conventional Treatment — Conventional rehabilitation
  Arms: Conventional Group (GC)

SUMMARY:
The performance of activities of daily living (ADL) depends to a large extent on the functionality of the upper limb and hand. Stroke is the leading cause of disability worldwide, with a significant individual, family and economic impact. After a stroke event, however, a large percentage of affected patients have a deficit of the hand and, six months after the acute event, 65% of patients with a deficit of the hand are unable to use and integrate the affected hand in activities of daily living, significantly reducing its quality. The impairment of strength, grip and general hand function makes it difficult to perform ADLs and affects the independence of functional activities, making the recovery of hand function an extremely challenging field in stroke rehabilitation.

DETAILED DESCRIPTION:
Rehabilitation of the hand in stroke patients has changed substantially over the last decades, with an increasing interest in the use of robotic devices for the treatment of the upper limb. Indeed, the use of such systems makes it possible to increase the amount and intensity of therapy, to standardise treatment, to provide complex but controlled multisensory stimulation, and to support the patient while performing various tasks, preventing inappropriate movements. Moreover, through robotic systems it is possible to acquire kinematic and kinetic data that are processed to obtain quantitative indices in order to objectively evaluate the patient's motor performance before and after the rehabilitation treatment.

Amadeo® (Tyromotion, Austria) is an end-effector type robotic device, specifically designed for hand treatment, effective in reducing hand disability in stroke patients.

The aim of the study is to evaluate the effects of robotic rehabilitation with an Amadeo® hand end-effector robot (Tyromotion, Austria):

(i) in terms of improved hand function (assessed by clinical and instrumental scales); (ii) on fatigue and quality of life. 24 patients will be recruited at the UOS Post-Acute Rehabilitation, Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome. Patients will be divided into two groups by randomization: one group (experimental group, GA) will perform specific rehabilitation for balance disorders using the end-effector robot Amadeo® (Tyromotion, Austria) 3 times a week, for 4 weeks (12 total sessions), for 45 minutes of treatment, in addition to the conventional treatment, and one group will perform only the conventional treatment (conventional group, GC), as a daily routine, as described below.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischaemic or haemorrhagic stroke documented by neuroimaging techniques (magnetic resonance imaging or computed tomography)
* Latency since acute event between 1 and 6 months;
* Cognitive ability to execute simple orders and understand the physiotherapist's instructions, assessed by Token Test (score ≥ 26.5);
* Ability to understand and sign informed consent.

Exclusion Criteria:

* Presence of a pincer grip "possible against resistance but weaker than the contralateral" as assessed by the Upper Limb Motricity Index ≥ 26;
* Behavioural, cognitive disorders and/or reduced compliance that could interfere with rehabilitation treatment;
* Presence of ankylosis as assessed by the modified Ashworth Scale ≥ 4;
* Inability to discriminate distinctly between images displayed on a monitor placed at eye level of each subject at a distance of approximately 50 cm, even with corrective glasses;
* Inability to provide informed consent.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment - Upper Extremity (FMA-UE) | Change from Baseline FMA-UE at 4 weeks
  The Fugl-Meyer Assessment - Upper Extremity (FMA-UE) is a stroke-specific, performance-based impairment index. Upper Extremity section is designed to assess motor functioning, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment.
  For each item, a score can be assigned on direct observation of performance. The scale items are scored according to the ability to complete the item using a 3-point ordinal scale where 0=not able to perform, 1=performs partially and 2=performs completely.
  The motor function macro-area has a maximum total score of 66; the sensitivity macro-area has a maximum total score of 60.

SECONDARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) | Change from Baseline MFIS at 4 weeks
  The MFIS is an instrument that provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The full-length MFIS consists of 21 items while the abbreviated version has 5 items. The MFIS is a structured, self-report questionnaire that the patient can generally complete with little or no intervention from an interviewer. However, patients with visual or upper extremity impairments may need to have the MFIS administered as an interview. Interviewers should be trained in basic interviewing skills and in the use of this instrument.
  The total score for the MFIS is the sum of the scores for the 21 items. Individual subscale scores for physical, cognitive, and psychosocial functioning can also be generated by calculating the sum of specific sets of items.
Fatigue Scale for Motor and Cognitive Function (FSMC) | Change from Baseline FSMC at 4 weeks
  The FSMC is an assessment of MS-related cognitive and motor fatigue. A Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question. Thus minimum value is 20 (no fatigue at all) and maximum value is 100 (severest grade of fatigue). Two subscales (mental and physical fatigue) can be made. Items included in the subscale mental are 1-4-7-8-11-13-15-17-18-20 and items included in the subscale physical are 2-3-5-6-9-10-12-14-16-19.
The Medical Research Council (MRC) Scale | Change from Baseline MRC at 4 weeks
  The MRC Scale is a 6-value scale for measuring strength through the observation of movement and muscle behaviour for grades 0 to 3 and the administration of Manual Muscle Tests for grades 4 and 5.
  The MRC Scale provides a score ranging from 0 to 5:
  0 Absence of contraction
  1. Hint of muscle contraction
  2. Active movement that eliminates the force of gravity
  3. Active movement against the force of gravity
  4. Active movement against the force of gravity and a resistance
  5. Normal force
Motricity Index - Upper Limb (MI-UL) | Change from Baseline MI-UL at 4 weeks
  MI-UL can be used to assess the upper limb motor impairment in a patient who has had a stroke.
  Test for each upper limb:
  pincer grip elbow flexion shoulder abduction For the pincer grip: 0 points, no movement 19 points, grip possible but not against gravity 33 points, normal grip For all other items: 0 points, no movement 14 points, Visible movement but not for the entire joint range or against gravity 19 points, movement possible for the entire joint range against gravity but not against resistance 33 points movement performed with normal force Each segment has a total score obtained by adding the value "1" to the score of each individual item. The total score then ranges from 1 (no movement) to 100 (normal movement).
Stroke Upper Limb Capacity Scale (SULCS) | Change from Baseline SULCS at 4 weeks
  The SULCS is a scale that assesses various arm and hand skills in the hemiplegic patient; in particular, it assesses highly functional movements related to activities of daily living.
  It consists of 10 items, assessable with a score of 0 or 1 (not performed/executed correctly), of which 3 items for limb skills without hand activity 4 items for limb skills and simple hand skills 3 items for complex hand skills The SULCS is a hierarchical scale: if the patient has poor upper limb skills and is unable to perform 3 consecutive items, all subsequent items will automatically receive a score of 0 without having to be performed.
  The maximum scale score is 10.
9-Hole Peg test (9HPT) | Change from Baseline 9HPT at 4 weeks
  The 9HPT is used to measure finger dexterity. The patient is asked to take the pegs from a container, one by one, and insert them into the holes in the board, as quickly as possible, using only his hand to assess. He/she must then remove them, one at a time, and reinsert them into the container.
  The final score is given by the time it takes the patient to complete the test.
Box&Block test (BBT) | Change from Baseline BBT at 4 weeks
  The BBT) measures unilateral gross manual dexterity. It is a quick, simple and inexpensive test.
  The BBT consists of a wooden box divided into two compartments by a divider and 150 blocks. The administration of the BBT consists of asking the patient to move, one at a time, the maximum number of blocks from one compartment of the box to another of equal size, within 60 seconds. The test must begin with the upper limb unaffected.
  The score is given according to the number of blocks moved from one compartment to another in 60 seconds. The score is assigned to each hand separately. Higher scores indicate better manual dexterity.
Modified Ashworth Scale (MAS) | Change from Baseline MAS at 4 weeks
  It is performed by first extending the patient's limb from a position of maximum possible flexion to maximum possible extension.
  The score ranges from 0 to 4:
  0 No increase in tone
  1 Slight increase in tone, giving a signal when there is a slight increase in muscle tone, manifested when the limb is moved into flexion or extension.
  1+ slight increase in muscle tone, manifested by a jerk followed by minimal resistance throughout the movement (ROM) 2 more marked increase in tone, but more marked increase in muscle tone through most of the limb easily flexed 3 marked increase in tone, difficult passive movement 4 stiff limb in flexion or extension
HandGrip Test (HGT) | Change from Baseline HGT at 4 weeks
  HGT is a test performed with a dynamometer, which goes to assess muscle strength (in kilograms). Starting with the elbow flexed to 90°, the patient must squeeze the dynamometer as hard as they can at one time. Three repeated measurements are taken on each side 20 seconds apart.
  The average of the three assessments is used as the final value.
modified Barthel Index (mBI) | Change from Baseline mBI at 4 weeks
  mBI for activities of daily living is meant to be used in the assessment of patient performance (or degree of assistance required) with respect to self-care, sphincter management, transfers and locomotion. The index consist of 10 items (each scored with a number of points) that relate to activities of daily living (ADLs) where the final score is calculated by summing the points awarded to each item. A five-point rating scales for each item to improve sensitivity to detecting change.
  The 10 items assessed relate to:
  Help needed with feeding; Help needed with bathing; Help needed with grooming; Help needed with dressing; Presence or absence of fecal incontinence; Presence or absence of urinary incontinence; Help needed with transfers; Help needed with walking; Help needed with climbing stairs.
  Interpretation:
  91-100 Slight dependency 61-90 Moderate dependency 21-60 Severe dependency 0-20 Total dependency
EuroQol- 5 Dimension (EQ-5D) | Change from Baseline EQ-5D at 4 weeks
  EQ-5D is an instrument which evaluates the generic quality of life. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ- 5D index an utility scores anchored at 0 for death and 1 for perfect health.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Giovannini, MD, phD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy